CLINICAL TRIAL: NCT01708174
Title: A Phase II, Multi-center, Open-label, Single-arm Study of the Efficacy and Safety of Oral LDE225 in Patients With Hh-pathway Activated Relapsed Medulloblastoma
Brief Title: A Phase II Study of Oral LDE225 in Patients With Hedge-Hog (Hh)-Pathway Activated Relapsed Medulloblastoma (MB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225C2301
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Medulloblastoma
Keywords: medulloblastoma,; relapsed,; pediatric,; children,; adults,; Hh pathway inhibitor,; LDE225
MeSH Terms: conditions — Medulloblastoma; Recurrence | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sonidegib (LDE225) (Experimental): 600 mg orally for adults and 500 mg/m2 orally for children
  Interventions: Drug: LDE225
- Temozolamide (TMZ) (Active Comparator): 150 to 200 mg/m2 for 5 sequential days every 4 weeks according to prescribing information until the study was amended to a single arm study.
  Interventions: Drug: TMZ

INTERVENTIONS:
Drug: LDE225 — Sonidegib for oral suspension was supplied in amber glass bottles. Sonidegib oral suspension was combined with the supplied reconstitution vehicle to a final concentration of 50 mg/mL.
  Arms: Sonidegib (LDE225)
Drug: TMZ — Temozolomide capsules were obtained locally by the Investigator
  Arms: Temozolamide (TMZ)

SUMMARY:
This Phase II study evaluated the safety and efficacy of LDE225 in adult and pediatric patients with Hh-pathway activated, relapsed MB.

DETAILED DESCRIPTION:
This study was a single-arm study of the efficacy and safety of oral sonidegib in patients with Hh-pathway activated relapsed medulloblastoma. It was initially designed as a randomized, controlled, open-label phase III study of adults and children with Hh-pathway activated MB whose disease had failed standard of care therapy, including radiation therapy (RT). The original study consisted of a randomized controlled part and a non-randomized uncontrolled part. Approximately 69 patients were to be randomized in a 2:1 ratio to receive sonidegib oral suspension or the active control, temozolomide (TMZ) capsules. Randomization was to be stratified according to age, <18 years versus ≥ 18 years. Approximately 40 patients were to receive sonidegib in the non-randomized uncontrolled part of the study. Following the enrollment of 11 patients, the study was amended to become a phase II single-arm study with only sonidegib, and the target enrollment was changed to 20 patients. Prior to the study amendment, TMZ participants whose disease progressed while on TMZ were permitted to crossover to sonidegib. After the amendment, participants receiving TMZ were crossed over to sonidegib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of MB, who have experienced relapse or progression after standard-of-care therapy including radiotherapy. Patients currently receiving steroids must have been on a stable (or decreasing) dose for at least 5 days before initiating study therapy.
* Only patients with a test result, using the 5-gene Hh signature assay, indicating Hhpathway activated MB are eligible for this study. All available tumor material obtained at any time during the course of the patient's disease should be submitted for these analyses
* At least one measurable lesion defined as lesion(s) that can be accurately measured in at least two dimensions and is ≥ 10 mm in each dimension by Gadolinium (Gd)-MRI, irrespective of slice thickness/reconstruction interval, for CNS lesions and CT or MRI (with or without contrast) for non-CNS lesions. All patients with CNS lesions must have a brain MRI with and without gadolinium and a spine MRI with gadolinium within 2 weeks prior to first dose of study treatment.
* Performance Status corresponding to ECOG score of 0, 1, or 2:

  1. Karnofsky performance status score ≥ 50 for patients >16 years of age
  2. Lansky performance status score ≥ 50 for patients ≤ 16 years of age
* Adequate bone marrow function as defined as:

  1. Peripheral absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  2. Platelet count ≥ 80 x 109/L
  3. Hemoglobin (Hgb) ≥ 9 g/dL
* Serum CK ≤1.5 ULN

Exclusion Criteria:

* Prior treatment with a Smoothened inhibitor Systemic anticancer treatment within 2 weeks before first dose of study treatment (6 weeks for nitrosourea, mitomycin, and monoclonal antibodies).
* Focal radiation therapy within 4 weeks before first dose of study treatment, or full spinal radiotherapy within 3 months before first dose of study treatment.
* Patients who have neuromuscular disorders that are associated with elevated CK (eg, inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Patients receiving treatment with medications that are known to be strong inhibitors or inducers of CYP3A4/5 or are metabolized by CYP2B6 and CYP2C9, that have narrow therapeutic indices that cannot be discontinued at least 2 weeks before first dose of study treatment and for the duration of the study
* Patients receiving unstable or increasing doses of corticosteroids. If patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms, dose must have been stabilized (or decreasing) for at least 5 days before first dose of study treatment.

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (8):
  - Ann & Robert H. Lurie Children Dept of Oncology, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins Med. Dept Onc, Baltimore, Maryland
  - Dana Farber Cancer Institute SC-7, Boston, Massachusetts
  - Columbia University Medical Center- New York Presbyterian Dept of Oncology, New York, New York
  - Cincinnati Children's Hospital Medical Center Division of Hema/Onco., Cincinnati, Ohio
  - Children's Hospital of Pittsburgh Dept of Oncology, Pittsburgh, Pennsylvania
  - University of Texas/MD Anderson Cancer Center SC-3, Houston, Texas
  - Seattle Cancer Care Alliance Dept Oncology, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Perth, Western Australia
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (7):
  - Novartis Investigative Site, Bordeaux, Aquitaine
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
- Italy (4):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia, Russia
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Esplugues de Llobregat, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Gothenburg, Sweden
- Novartis Investigative Site, Zurich, Switzerland
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Leeds

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analyses were performed by treatment and by age group.
Groups:
- Sonidegib (LDE225) Children: 500 mg/m2 orally
- Sonidegib (LDE225) Adults: 600 mg orally
- Temozolomide (TMZ): 150 to 200 mg/m2 for 5 sequential days every 4 weeks according to prescribing information until the study was amended to a single arm study.
Period: Treatment Period
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Started | 2 | 16 | 4
Pharmacokinetic Analysis Set | 2 | 13 | 0
Completed | 1 | 14 | 3
Not Completed | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Period: Survival Follow-up
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Started | 1 | 10 | 0
Completed | 1 | 10 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ) | Total
Number analyzed (Participants) | 2 | 16 | 4 | 22
Age, Continuous [Median (Full Range); unit: Years] | 8.5 (6.36) [4.0 to 13.0] | 37.0 (8.17) [24.0 to 51.0] | 35.5 (3.16) [31.0 to 38.0] | 35.0 (10.73) [4.0 to 51.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 9
  Male | 0 | 11 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR) According to Independent Review Committee (IRC) From Date First Participant Randomized, 13-Sep-2013 to Date of Data Cut-off, 15-Nov-2016
Description: ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) (as per tumor response guidelines and criteria for Medulloblastoma). The IRC evaluated all radiological images and applicable clinical data (i.e., neurological examination, steroid use and cerebrospinal fluid (CSF) results as applicable). Assessments after crossover were not included for TMZ participants.
Time Frame: from date first participant randomized, 13-Sep-2013 to date of data cut-off, 15-Nov-2016
Population: The full analysis set (FAS) was analyzed. The FAS included all randomized and non-randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Number analyzed (Participants) | 2 | 16 | 4
Percentage of participants | 0.0 | 18.8 | 0.0

2. Secondary Outcome: Progression Free Survival (PFS) According to IRC From Date First Participant Randomized, 13-Sep-2013 to Date of Data Cut-off, 15-Nov-2016
Description: PFS was defined as the time from date of randomization to the date of event defined as the first documented progression or death due to any cause (as per tumor response guidelines and criteria for Medulloblastoma). The IRC evaluated all radiological images and applicable clinical data (i.e., neurological examination, steroid use and cerebrospinal fluid (CSF) results as applicable). TMZ participants without event prior to crossover were censored.
Time Frame: from date first participant randomized, 13-Sep-2013 to date of data cut-off, 15-Nov-2016
Population: The FAS was analyzed. The FAS included all randomized and non-randomized participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Number analyzed (Participants) | 2 | 16 | 4
months | 1.6 [NA to NA] — The lower and upper 95% confidence intervals (CI) were not estimable because there were only 2 participants analyzed. With only 2 participants, it is not uncommon to have 'not estimable' for the limits. | 3.3 [1.7 to 17.1] | 2.9 [0.9 to 4.0]

3. Secondary Outcome: PFS According to Local Investigator Assessment From Date First Participant Randomized, 13-Sep-2013 to Date of Data Cut-off, 15-Nov-2016
Description: PFS was defined as the time from date of randomization to the date of event defined as the first documented progression or death due to any cause. PFS was evaluated by local Investigator assessment per tumor response guidelines and criteria for Medulloblastoma.
Time Frame: from date first participant randomized, 13-Sep-2013 to date of data cut-off, 15-Nov-2016
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Number analyzed (Participants) | 2 | 16 | 4
months | NA [1.6 to NA] — The median and upper limit of the 95% confidence interval were not estimable because there were too few events. | 3.3 [1.6 to 13.0] | 2.9 [0.9 to 4.0]

4. Secondary Outcome: Percentage of Participants With ORR According to Local Investigator Assessment From Date First Participant Randomized, 13-Sep-2013 to Date of Data Cut-off, 15-Nov-2016
Description: ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR). ORR was evaluated by local Investigator assessment per tumor response guidelines and criteria for Medulloblastoma. Assessments after crossover were not included for TMZ patients.
Time Frame: from date first participant randomized, 13-Sep-2013 to date of data cut-off, 15-Nov-2016
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Number analyzed (Participants) | 2 | 16 | 4
Percentage of participants | 0.0 | 25.0 | 0.0

5. Secondary Outcome: Duration of Response (DoR) According to Local Investigator Assessment From Date First Participant Randomized, 13-Sep-2013 to Date of Data Cut-off, 15-Nov-2016
Description: DoR was defined as the time from the first documented onset of confirmed PR or CR to the date of PD/relapse or death due to medulloblastoma. DoR was evaluated by local Investigator assessment per tumor response guidelines and criteria for Medulloblastoma. TMZ participants without an event prior to crossover were censored.
Time Frame: from date first participant randomized, 13-Sep-2013 to date of data cut-off, 15-Nov-2016
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Number analyzed (Participants) | 2 | 16 | 4
months | NA [NA to NA] — The median and lower and upper 95% CI could not be calculated because there were too few events. | 8.5 [4.1 to 16.6] | NA [NA to NA] — The median and lower and upper 95% CI could not be calculated because there were too few events.

6. Secondary Outcome: Overall Survival (OS) From Date First Participant Randomized, 13-Sep-2013 to Date of Data Cut-off, 15-Nov-2016
Description: OS was defined as the time from date of randomization to date of death due to any cause. All deaths are considered, including deaths occurred after crossover for TMZ participants.
Time Frame: from date first participant randomized, 13-Sep-2013 to date of data cut-off, 15-Nov-2016
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Temozolomide (TMZ)
Number analyzed (Participants) | 2 | 16 | 4
months | NA [4.5 to NA] — The median and upper 95% CI could not be calculated because there were too few events. | 9.5 [4.9 to 15.6] | NA [1.2 to NA] — The median and upper 95% CI could not be calculated because there were too few events.

7. Secondary Outcome: Pharmacokinetics (PK): Summary of Plasma Trough Concentrations for Sonidegib (LDE225)
Description: Blood samples were collected for assessment. The children's group was analyzed up until week 25 only.
Time Frame: Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49 and 53
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults
Number analyzed (Participants) | 2 | 13
ng/mL
  Week 1 (n=2,11) | 0.00 (0.00) | 0.00 (0.00)
  Week 3 (n=2,10) | 2890 (1240) | 761 (519)
  Week 5 (n=2,8) | 4930 (1380) | 1090 (700)
  Week 7 (n=1,8) | 2810 (NA) — Standard deviation (SD) does not apply when n=1. | 1450 (842)
  Week 9 (n=1,8) | 4670 (NA) — SD does not apply when n=1. | 1530 (682)
  Week 13 (n=1,4) | 3680 (NA) — SD does not apply when n=1. | 2330 (1100)
  Week 17 (n=1,6) | 3060 (NA) — SD does not apply when n=1. | 1880 (730)
  Week 21 (n=1,5) | 3770 (NA) — SD does not apply when n=1. | 2270 (915)
  Week 25 (n=1,4) | 1890 (NA) — SD does not apply when n=1. | 2050 (625)
  Week 29 (n=NA,4) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2050 (906)
  Week 33 (n=NA,4) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2180 (512)
  Week 37 (n=NA,3) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2850 (306)
  Week 41 (n=NA,4) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2370 (916)
  Week 45 (n=NA,2) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2890 (290)
  Week 49 (n=NA,2) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2330 (990)
  Week 53 (n=NA,2) | NA (NA) — PK analysis for the Children group was done up until week 25 only. | 2080 (764)

ADVERSE EVENTS:
Groups:
- Sonidegib (Total): Sonidegib (Total)
Arm/Group | Sonidegib (LDE225) Children | Sonidegib (LDE225) Adults | Sonidegib (Total) | Temozolomide (TMZ)
Serious Adverse Events (participants affected / at risk) | 2/2 | 9/16 | 11/18 | 1/4
Other Adverse Events (participants affected / at risk) | 2/2 | 16/16 | 18/18 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sonidegib (LDE225) Children (N=2) | Sonidegib (LDE225) Adults (N=16) | Sonidegib (Total) (N=18) | Temozolomide (TMZ) (N=4)
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 2 | 2 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 1 | 0
PAIN (General disorders) | 0 | 1 | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1 | 1 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 2 | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
SEIZURE (Nervous system disorders) | 0 | 1 | 1 | 0
THROMBOSIS IN DEVICE (Product Issues) | 1 | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 1 | 0
DRUG DEPENDENCE (Psychiatric disorders) | 0 | 1 | 1 | 0
HALLUCINATION (Psychiatric disorders) | 0 | 1 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
EMBOLISM (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sonidegib (LDE225) Children (N=2) | Sonidegib (LDE225) Adults (N=16) | Sonidegib (Total) (N=18) | Temozolomide (TMZ) (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 1 | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 2 | 2 | 0
EAR CONGESTION (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
DIABETES INSIPIDUS (Endocrine disorders) | 0 | 1 | 1 | 0
DIPLOPIA (Eye disorders) | 0 | 1 | 1 | 0
PHOTOPHOBIA (Eye disorders) | 0 | 1 | 1 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 2 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 1 | 0
AEROPHAGIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 6 | 6 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 3 | 4 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 5 | 5 | 3
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 1 | 1 | 0
REGURGITATION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
TOOTH DISCOLOURATION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
TOOTH LOSS (Gastrointestinal disorders) | 0 | 1 | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 7 | 9 | 1
ASTHENIA (General disorders) | 0 | 2 | 2 | 1
FATIGUE (General disorders) | 0 | 7 | 7 | 2
GAIT DISTURBANCE (General disorders) | 0 | 1 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 2 | 2 | 1
PAIN (General disorders) | 0 | 2 | 2 | 0
PYREXIA (General disorders) | 0 | 2 | 2 | 0
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 1 | 1 | 0
ACINETOBACTER INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
FOLLICULITIS (Infections and infestations) | 0 | 2 | 2 | 0
ORAL HERPES (Infections and infestations) | 1 | 0 | 1 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 4 | 4 | 0
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 1 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 | 3 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 2 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 1 | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 7 | 8 | 1
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 1 | 1 | 2 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 3 | 3 | 0
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 | 1 | 1 | 0
BODY TEMPERATURE INCREASED (Investigations) | 0 | 1 | 1 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 1 | 1 | 0
CRYSTAL URINE PRESENT (Investigations) | 0 | 1 | 1 | 0
GRANULOCYTE COUNT INCREASED (Investigations) | 0 | 1 | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 5 | 5 | 1
OXYGEN SATURATION DECREASED (Investigations) | 0 | 1 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 1 | 1 | 1
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 1 | 1 | 0
RED BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 1 | 0
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 0 | 1 | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 2 | 2 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 4 | 4 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 3 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 4 | 4 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 3 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1
APHASIA (Nervous system disorders) | 0 | 2 | 2 | 0
ATAXIA (Nervous system disorders) | 0 | 1 | 1 | 1
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 0 | 0 | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 3 | 3 | 1
DROOLING (Nervous system disorders) | 0 | 1 | 1 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 1 | 1 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 5 | 5 | 0
FACIAL NERVE DISORDER (Nervous system disorders) | 0 | 1 | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 3 | 5 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 1 | 1 | 0
IIIRD NERVE DISORDER (Nervous system disorders) | 0 | 1 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 1 | 1 | 0
MUSCLE SPASTICITY (Nervous system disorders) | 1 | 1 | 2 | 0
MYOCLONUS (Nervous system disorders) | 0 | 1 | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 2 | 2 | 0
NYSTAGMUS (Nervous system disorders) | 0 | 1 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 1 | 1 | 0
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 0 | 1 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 3 | 3 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 2 | 2 | 0
DELIRIUM (Psychiatric disorders) | 0 | 2 | 2 | 0
DEPRESSION (Psychiatric disorders) | 0 | 2 | 2 | 0
INSOMNIA (Psychiatric disorders) | 0 | 3 | 3 | 0
IRRITABILITY (Psychiatric disorders) | 0 | 1 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 1 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 1 | 0
APNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 6 | 8 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 1 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 2 | 2 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.